CLINICAL TRIAL: NCT05074888
Title: A Multicenter, Double-blind, Placebo-controlled, Parallel-group, Randomized Clinical Trial of Efficacy and Safety of Prospekta in the Treatment of Patients With Post-COVID-19 Asthenia.
Brief Title: Сlinical Trial of Efficacy and Safety of Prospekta in the Treatment of Post-COVID-19 Asthenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-MAP-006
Record Dates: First submitted 2021-10-05; First posted 2021-10-12 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-01

CONDITIONS: Post-acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, parallel-group, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospekta (Experimental): Tablet for oral use. 1 tablet twice daily. The tablets are taken outside of meals (between meals or 15 minutes before eating or drinking), keep the tablets in the mouth, without swallowing, until completely dissolved.
  Interventions: Drug: Prospekta
- Placebo (Placebo Comparator): Tablet for oral use. Placebo using Prospekta scheme.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prospekta — Oral administration.
  Arms: Prospekta
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
The multicenter, double-blind, placebo-controlled, parallel-group, randomized clinical trial.

The objective of this study is to evaluate the efficacy and safety of Prospekta in the treatment of asthenia in patients after the coronavirus infectious disease (COVID-19).

DETAILED DESCRIPTION:
Design: the multicenter, double-blind, placebo-controlled, parallel-group, randomized clinical trial.

The study will enroll adult patients of either gender aged 18 to 65 years after new coronavirus infection of 2019 (COVID-19) with symptoms of asthenia that appeared during or after an acute coronavirus infection (COVID-19) and persisting 4 to 12 weeks from the onset of coronavirus infection.

After the patient signs the patient information sheet and the informed consent form for participation in the study, complaints, medical history, physical examination, registration of vital signs are collected, the patient fills in the Fatigue Severity Scale (FSS) and Hospital Anxiety and Depression Scale (HADS). A six-minute walk test (6MWT) is carried out. The physician evaluates the severity of asthenia with FSS scale and records concomitant medications, co-morbidities and concurrent conditions.

If a patient meets all inclusion criteria and does not have any of the exclusion criteria at Visit 1 (Day 1), he/she is randomized to one of two groups: Group 1 - patients receive Prospekta at a dose of 1 tablet twice daily for 4 weeks; Group 2 - patients receive placebo on the study drug regimen.

The trial will use electronic patient diaries (EPD). The patient should record any possible deterioration (if applicable) in the EPD. At Visit 1 (Day 1), the physician will provide guidance on how to work with EPD, so that the patient can use it independently in the future.

At Visit 2 (Week 4 ± 3 days), the physician will collect patient's complaints, record physical examination data and vital signs as well as any changes in concurrent diseases and conditions. The patient fills out the FSS and HADS scales. A 6MWT is carried out. The physician monitors the prescribed treatment and use of concomitant medications, evaluates the safety of the study treatment and patient's compliance, filling out the diary.

The patient stops taking the study drug. At the end of the study treatment period, the patient is monitored for 4 weeks (follow-up period).

At Visit 3 (final visit, Week 8 ± 3 days), the physician collects patient's complaints, records physical examination data and vital signs, changes in concomitant diseases and conditions. The patient fills in the FSS and HADS scales. A 6MWT is carried out. The physician evaluates the safety of the study treatment, checks the completion of the diary.

During the study the patients are allowed to take medications for their chronic conditions, except for medicines listed as "Prohibited concomitant treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Adults of either gender aged 18 to 65 years inclusive.
2. Patients within 4-12 weeks of the confirmed COVID-19 onset .
3. Symptoms of asthenia that appeared during or after an acute new coronavirus infection (COVID-19), persisting from 4 to 12 weeks from the onset of coronavirus infection.
4. Presence of asthenia (≥36 on the FSS scale).
5. Patients who agreed to use a reliable method of contraception during the study (for men and women with reproductive potential).
6. Presence of a signed information sheet and informed consent form for participation in a clinical trial.

Exclusion Criteria:

1. History / suspicion of cancer of any localization (with the exception of benign neoplasms).
2. More than 75% of lung tissue damage during the period of COVID-19 disease (CT 4).
3. Cerebrovascular diseases with the development of moderate to severe cognitive impairments.
4. Uncontrolled arterial hypertension characterized by the following blood tension values: systolic blood pressure > 180 mm Hg and/or diastolic blood pressure > 110 mm Hg.
5. Myocardial infarction, stroke in the previous 6 months.
6. Nervous system disorders with persistent neurological impairment.
7. Autoimmune diseases.
8. Decompensated diseases of the cardiovascular system, liver, kidney, gastrointestinal tract, and metabolic, respiratory, endocrine or hematological diseases, peripheral vascular disorders.
9. Any severe comorbidity which, in the opinion of the investigator, may affect patient participation in the clinical trial.
10. Hypersensitivity to any of the components of the study drug.
11. Hereditary lactose intolerance, lactose malabsorption, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
12. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial (for men and women with reproductive potential).
13. Patients, who, from the investigator's point of view, will not comply with study observation requirements or study drug administration procedures..
14. Prior history of mental illness, alcoholism or drug abuse, that the investigator's opinion, will interfere with successful study procedures.
15. Use of any medications listed in "Prohibited concomitant treatment" within 1 week before enrollment.
16. Participation in other clinical studies within 3 months prior to enrollment in the study.
17. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. "Immediate relative" means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
18. Participants who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- Russia (32):
  - Belgorod Regional Clinical Hospital of St. Joasaph, Belgorod
  - Clinical hospital "RZD-Medicine" of Chelyabinsk city, Chelyabinsk
  - Ivanovo clinical hospital named after Kuvaevs/Polyclinic #10, Ivanovo
  - City Clinical Hospital # 9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Kazan State Medical University, Department of Propedeutics of Internal Diseases named after prof. S.S. Zimnitsky, Kazan'
  - Kazan State Medical University, Kazan'
  - Kirov State Medical University, Hospital Therapy Department, Kirov
  - Kuban State Medical University, Infectious Diseases and Phthisiopulmonology, Krasnodar
  - Krasnogorsk city hospital #r 1, Krasnogorsk
  - City Clinical Hospital named after V.M. Buyanov of the Moscow City Health Department, Moscow
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Llc "Verum Medical", Moscow
  - Moscow State Medical and Dental University named after A.I. Evdokimov, Department of Faculty Therapy and Occupational Diseases, Moscow
  - Nizhny Novgorod Research Institute of Hygiene and Occupational Pathology, Nizhny Novgorod
  - Llc "Nizhmedklinika", Nizhny Novgorod
  - City Emergency Hospital of Rostov-on-Don, Rostov-on-Don
  - Ryazan State Medical University named after acad. I.P. Pavlov, Department of Outpatient Therapy and Preventive Medicine, Ryazan
  - Llc "Ava-Peter", Saint Petersburg
  - LLC "Energy of Health", Saint Petersburg
  - LLC Medical center" Reavita Med SPb ", Saint Petersburg
  - City polyclinic # 51, Saint Petersburg
  - City Polyclinic # 34, Saint Petersburg
  - Saratov State Medical University named after V. I. Razumovsky, Neurology Department named after K.N. Tretyakov, Saratov
  - LLC "Scientific Medical Center for General Therapy and Pharmacology", Stavropol
  - Bashkir State Medical University, Internal Medicine Department, Ufa
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Vsevolozhsk clinical interdistrict hospital, Vsevolozhsk
  - LLC "Center for Medical Consulting and Research - PRACTICE", Yaroslavl
  - Clinical Hospital # 2, Yaroslavl
  - Clinical Hospital # 9, Yaroslavl
  - LLC "Family Clinic", Yekaterinburg
  - Central city hospital # 7, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospekta | Placebo
Started | 330 | 346
Completed | 330 | 346
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospekta | Placebo | Total
Number analyzed (Participants) | 330 | 346 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.5) | 42.8 (12.6) | 43.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 236 | 452
  Male | 114 | 110 | 224
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 330 | 346 | 676

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean FSS Score.
Description: Fatigue Severity Scale (FSS). Change in the mean FSS score after 4 weeks of treatment. The total score of the scale, which consists of 9 questions, varies between 9-63. This scale consists of a 7-point Likert scale. 1 point means strongly disagree, 7 means strongly agree. People are asked to mark the appropriate options for each question taking into account their status in the last 1 month period. A total of 36 points and above indicate fatigue. A higher score is indicated high level of fatigue.
Time Frame: after 4 weeks of treatment
Population: Six patients were excluded from the trial before 4 week therefore no data was collected on 4 weeks timepoint (3 patients from Prospekta group and 3 patients from Placebo group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 327 | 343
score on a scale
  Baseline | 46.4 (6.9) | 45.9 (6.6)
  After 4 weeks | 29.9 (9.2) | 31.9 (9.9)
  ∆ between baseline and 4 weeks later | 16.5 (9.5) | 14.0 (9.4)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 4 weeks later row; Test type: Superiority; p = 0.0016, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Distance of the 6-minute Walk Test.
Description: Change in distance when performing the 6-minute walk test after 4 weeks of treatment. The test is carried out with the aim of objectively assessing the patient's physical tolerance. The patient should walk the maximum possible distance for himself at his own pace on a flat surface in 6 minutes.
Time Frame: after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 328 | 343
meters
  Baseline | 426.4 (119.2) | 416.9 (112.8)
  After 4 weeks | 457.8 (118.2) | 444.7 (110.7)
  ∆ between baseline and 4 weeks later | 31.4 (44.5) | 27.8 (38.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 4 weeks later row; Test type: Superiority; p = 0.3183, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in the Severity of Anxiety on the HADS Subscale.
Description: Hospital Anxiety and Depression Scale (HADS). Change in the severity of anxiety and depression on the HADS subscales after 4 weeks of treatment. The scale is composed of 14 statements serving 2 subscales: "anxiety" (odd items - 1, 3, 5, 7, 9, 11, 13) and "depression" (even items - 2, 4, 6, 8, 10, 12 , 14). Each statement corresponds to 4 answer options, reflecting the gradation of the severity of the sign and coded according to the increase in the severity of the symptom from 0 (no) to 3 (maximum severity). When interpreting the results, the total indicator for each subscale is taken into account, while there are 3 areas of its values:
  0-7 - "norm" (absence of reliably expressed symptoms of anxiety and depression); 8-10 - "subclinical anxiety / depression"; 11 and above - "clinical anxiety / depression". The anxiety subscale ranges from 0 to 21, with higher values reflecting a worse outcome.
Time Frame: after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 326 | 343
score on a scale
  Baseline | 8.5 (4.1) | 8.8 (3.9)
  After 4 weeks | 5.5 (3.2) | 6.0 (3.3)
  ∆ between baseline and 4 weeks later | 3.0 (3.2) | 2.8 (3.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 4 weeks later row; Test type: Superiority; p = 0.5805, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in the Severity of Depression on the HADS Subscale.
Description: Hospital Anxiety and Depression Scale (HADS). Change in the severity of depression on the HADS subscale after 4 weeks of treatment. The scale is composed of 14 statements serving 2 subscales: "anxiety" (odd items - 1, 3, 5, 7, 9, 11, 13) and "depression" (even items - 2, 4, 6, 8, 10, 12 , 14). Each statement corresponds to 4 answer options, reflecting the gradation of the severity of the sign and coded according to the increase in the severity of the symptom from 0 (no) to 3 (maximum severity). When interpreting the results, the total indicator for each subscale is taken into account, while there are 3 areas of its values:
  0-7 - "norm" (absence of reliably expressed symptoms of anxiety and depression); 8-10 - "subclinical anxiety / depression"; 11 and above - "clinical anxiety / depression". The depression subscale ranges from 0 to 21, with higher values reflecting a worse outcome.
Time Frame: after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 327 | 343
score on a scale
  Baseline | 8.1 (3.7) | 8.3 (3.8)
  After 4 weeks | 4.7 (2.9) | 5.2 (3.0)
  ∆ between baseline and 4 weeks later | 3.4 (3.0) | 3.1 (3.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 4 weeks later row; Test type: Superiority; p = 0.2143, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in the Mean FSS Score Within Follow-up Period.
Description: Change in mean FSS score over 4 weeks of follow-up period at the end of treatment. The total score of the scale, which consists of 9 questions, varies between 9-63. This scale consists of a 7-point Likert scale. 1 point means strongly disagree, 7 means strongly agree. People are asked to mark the appropriate options for each question taking into account their status in the last 1 month period. A total of 36 points and above indicate fatigue. A higher score is indicated high level of fatigue.
Time Frame: after 4 weeks of treatment and after 4 weeks of follow-up at week 8
Population: One patient in Prospekta group was excluded from the trial before finishing follow-up period therefore no data was collected within 4 weeks of follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 327 | 343
score on a scale
  After 4 weeks | 29.9 (9.2) | 31.9 (9.9)
  After 8 weeks: number analyzed (Participants) | 326 | 343
  After 8 weeks | 22.9 (9.0) | 25.0 (10.2)
  ∆ between value after 4 weeks and after 8 weeks: number analyzed (Participants) | 326 | 343
  ∆ between value after 4 weeks and after 8 weeks | 7.1 (6.3) | 7.0 (6.9)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between value after 4 weeks and after 8 weeks row; Test type: Superiority; p = 0.8156, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Distance of the 6-minute Walk Test Within Follow-up Period.
Description: Change in distance when performing the 6-minute walk test over a 4-week follow-up period at the end of treatment. The test is carried out with the aim of objectively assessing the patient's physical tolerance. The patient should walk the maximum possible distance for himself at his own pace on a flat surface in 6 minutes.
Time Frame: after 4 weeks of treatment and after 4 weeks of follow-up at week 8
Population: One patient in Prospekta group and three patients in Placebo group were excluded from the trial before finishing follow-up period therefore no data was collected within 4 weeks of follow-up.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 328 | 343
meter
  After 4 weeks | 457.8 (118.2) | 444.7 (110.7)
  After 8 weeks: number analyzed (Participants) | 327 | 340
  After 8 weeks | 472.9 (116.5) | 462.7 (110.1)
  ∆ between value after 4 weeks and after 8 weeks: number analyzed (Participants) | 327 | 340
  ∆ between value after 4 weeks and after 8 weeks | 15.9 (32.1) | 18.8 (32.0)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between value after 4 weeks and after 8 weeks row; Test type: Superiority; p = 0.1049, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in the Severity of Anxiety on the HADS Subscales Within Follow-up Period.
Description: Change in the severity of anxiety on the HADS subscales over a 4-week follow-up period at the end of treatment. The scale is composed of 14 statements serving 2 subscales: "anxiety" (odd items - 1, 3, 5, 7, 9, 11, 13) and "depression" (even items - 2, 4, 6, 8, 10, 12 , 14). Each statement corresponds to 4 answer options, reflecting the gradation of the severity of the sign and coded according to the increase in the severity of the symptom from 0 (no) to 3 (maximum severity). When interpreting the results, the total indicator for each subscale is taken into account, while there are 3 areas of its values:
  0-7 - "norm" (absence of reliably expressed symptoms of anxiety and depression); 8-10 - "subclinical anxiety / depression"; 11 and above - "clinical anxiety / depression". The anxiety subscale ranges from 0 to 21, with higher values reflecting a worse outcome.
Time Frame: after 4 weeks of treatment and after 4 weeks of follow-up at week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 327 | 343
score on a scale
  After 4 weeks | 5.5 (3.2) | 6.0 (3.3)
  After 8 weeks: number analyzed (Participants) | 326 | 340
  After 8 weeks | 4.0 (2.8) | 4.4 (3.0)
  ∆ between value after 4 weeks and after 8 weeks: number analyzed (Participants) | 326 | 340
  ∆ between value after 4 weeks and after 8 weeks | 1.5 (2.3) | 1.6 (2.3)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between value after 4 weeks and after 8 weeks row; Test type: Superiority; p = 0.7260, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in the Severity of Depression on the HADS Subscales Within Follow-up Period.
Description: Change in the severity of depression on the HADS subscales over a 4-week follow-up period at the end of treatment.
  The scale is composed of 14 statements serving 2 subscales: "anxiety" (odd items - 1, 3, 5, 7, 9, 11, 13) and "depression" (even items - 2, 4, 6, 8, 10, 12 , 14). Each statement corresponds to 4 answer options, reflecting the gradation of the severity of the sign and coded according to the increase in the severity of the symptom from 0 (no) to 3 (maximum severity). When interpreting the results, the total indicator for each subscale is taken into account, while there are 3 areas of its values:
  0-7 - "norm" (absence of reliably expressed symptoms of anxiety and depression); 8-10 - "subclinical anxiety / depression"; 11 and above - "clinical anxiety / depression". The depression subscale ranges from 0 to 21, with higher values reflecting a worse outcome.
Time Frame: after 4 weeks of treatment and after 4 weeks of follow-up at week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 327 | 343
score on a scale
  After 4 weeks | 4.7 (2.9) | 5.2 (3.0)
  After 8 weeks: number analyzed (Participants) | 326 | 340
  After 8 weeks | 3.4 (2.6) | 3.7 (2.8)
  ∆ between value after 4 weeks and after 8 weeks: number analyzed (Participants) | 326 | 340
  ∆ between value after 4 weeks and after 8 weeks | 1.4 (2.1) | 1.5 (2.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between value after 4 weeks and after 8 weeks row; Test type: Superiority; p = 0.6808, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Changes in Vital Signs (Pulse Rate (Heart Rate)).
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: after 4 weeks of treatment and within 4 weeks of the follow-up period at the end of the treatment.
Population: Lower patient count is due to missing data on visits 2 and 3.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 330 | 346
beats per minute
  Visit 1: baseline | 73.0 (6.9) | 73.4 (6.9)
  Visit 2: after 4 weeks of treatment: number analyzed (Participants) | 328 | 343
  Visit 2: after 4 weeks of treatment | 71.8 (5.8) | 71.9 (5.6)
  Visit 3: after 4 weeks of follow-up at week 8: number analyzed (Participants) | 327 | 340
  Visit 3: after 4 weeks of follow-up at week 8 | 71.6 (5.3) | 71.4 (5.5)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.54, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction of pulse rate (heart rate) from Visit 1 to 3 between Prospekta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

10. Secondary Outcome: Changes in Vital Signs (Respiration Rate (Breathing Rate)).
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: after 4 weeks of treatment and within 4 weeks of the follow-up period at the end of the treatment (Visit 1: baseline, Visit 2: after 4 weeks of treatment, and Visit 3: after 4 weeks of follow-up at week 8)
Population: Lower patient count is due to missing data on visits 2 and 3.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 330 | 346
breaths per minute
  Visit 1 | 16.3 (1.3) | 16.4 (1.3)
  Visit 2: number analyzed (Participants) | 328 | 343
  Visit 2 | 16.2 (1.2) | 16.2 (1.2)
  Visit 3 | 16.2 (1.2) | 16.2 (1.2)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.49, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction of respiration rate (breathing rate) from Visit 1 to 3 between Prospekta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

11. Secondary Outcome: Changes in Vital Signs (Blood Pressure).
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: as for outcome 10
Population: Lower patient count is due to missing data on visits 2 and 3.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 330 | 346
mmHg
  SBP/Visit 1 | 121.3 (8.6) | 120.9 (8.3)
  SBP/Visit 2: number analyzed (Participants) | 328 | 343
  SBP/Visit 2 | 121.1 (8.4) | 120.6 (8.1)
  SBP/Visit 3: number analyzed (Participants) | 327 | 340
  SBP/Visit 3 | 121.1 (8.2) | 120.4 (7.4)
  DBP/Visit 1 | 75.8 (6.5) | 75.8 (6.5)
  DBP/Visit 2: number analyzed (Participants) | 328 | 343
  DBP/Visit 2 | 75.8 (6.3) | 75.9 (6.3)
  DBP/Visit 3: number analyzed (Participants) | 327 | 340
  DBP/Visit 3 | 76.0 (6.1) | 75.4 (5.9)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to SBP/Visit1, SBP/Visit2 and SBP/Visit3 rows; Test type: Superiority; p = 0.87, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction of systolic blood pressure from Visit 1 to 3 between Prospekta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction
Statistical Analysis 2: Comparison: Prospekta vs Placebo; This analysis applies to DBP/Visit1, DBP/Visit2 and DBP/Visit3 rows; Test type: Superiority; p = 0.22, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction of diastolic blood pressure from Visit 1 to 3 between Prospekta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

12. Secondary Outcome: Presence of Adverse Events (AEs).
Description: The number of participants with adverse events (AEs). Based on medical records.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 330 | 346
Participants | 20 | 20
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact

13. Secondary Outcome: The Severity of AEs.
Description: The intensity (severity) of adverse events. Based on medical records.
Time Frame: 8 weeks
Measure: Number; unit: number of AEs
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 20 | 20
number of AEs
  Mild | 13 | 15
  Moderate | 11 | 13
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact

14. Secondary Outcome: The Outcome of AEs.
Description: The outcome of adverse events. Based on medical records.
Time Frame: 8 weeks
Measure: Number; unit: number of AEs
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 20 | 20
number of AEs
  Recovery/resolution | 22 | 26
  No recovery/resolution | 2 | 0
  Unknown | 0 | 2
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.17, Fisher Exact

15. Secondary Outcome: AEs Causal Relationship to the Study Drug.
Description: The adverse events causal relationship to the study drug. Based on medical records.
Time Frame: 8 weeks
Measure: Number; unit: number of AEs
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 20 | 20
number of AEs
  No relation | 20 | 15
  Probable | 3 | 4
  Possible | 1 | 0
  Doubtful | 0 | 9
Statistical Analysis 1: Comparison: Prospekta vs Placebo; Test type: Superiority; p = 0.004, Fisher Exact

ADVERSE EVENTS:
Time Frame: Reporting of AEs begins after the first dose of IP, continues throughout the study treatment period, and for 4 weeks after the last dose of IP during the follow-up period, up to 8 weeks.
Arm/Group | Prospekta | Placebo
All-Cause Mortality (participants affected / at risk) | 0/330 | 0/346
Serious Adverse Events (participants affected / at risk) | 0/330 | 0/346
Other Adverse Events (participants affected / at risk) | 20/330 | 20/346
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospekta (N=330) | Placebo (N=346)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Viral infection of the respiratory tract (Infections and infestations) | 2 (2) | 1 (1)
Herpes (Infections and infestations) | 0 (0) | 1 (1)
Laboratory confirmed coronavirus infection COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Acute respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Acute rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
BP above normal (Investigations) | 1 (1) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Lumbar spine pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dorsopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Root lumbar pain (Nervous system disorders) | 0 (0) | 1 (1)
Upper limb numbness (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disorder (Nervous system disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 2 (2) | 0 (0)
Cephalalgia (Nervous system disorders) | 0 (0) | 1 (1)
Ovarian hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Worsening of hypertension (Vascular disorders) | 2 (2) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Precardial pain (General disorders) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 1 (1)
Residual taste after drug administration (Product Issues) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
Tearfulness (Psychiatric disorders) | 1 (1) | 0 (0)
Back contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT05074888/Prot_SAP_000.pdf